CLINICAL TRIAL: NCT04204928
Title: Pre-Approval Access Program (PAAP) for Pralsetinib (BLU-667) in Patients With Unresectable or Metastatic NSCLC or MTC
Status: Approved for marketing | Type: Expanded Access
Sponsor: Blueprint Medicines Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: BLU-667-PAAP-01
Record Dates: First submitted 2019-12-17; First posted 2019-12-19 (Actual); Last update posted 2021-08-13 (Actual); Status verified 2021-08

CONDITIONS: Non-Small Cell Lung Cancer; Medullary Thyroid Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Carcinoma, Medullary | interventions — pralsetinib

STUDY DESIGN:
Expanded Access Types: Individual, Treatment

INTERVENTIONS:
Drug: pralsetinib (BLU-667) — Pralsetinib will be administered orally (PO) at a dose of 400 mg once daily (QD) in continuous 28 day cycles

SUMMARY:
This is a global, multicenter, open-label pre-approval access program to provide access to pralsetinib (BLU-667) until such time that pralsetinib becomes available through other mechanisms or the Sponsor chooses to discontinue the program.

ELIGIBILITY:
Inclusion Criteria:

1a. Pathologically documented and definitively diagnosed non-resectable or metastatic NSCLC with a RET fusion for patients who are either treatment naïve, or who have been previously treated with systemic therapy. In the presence of a primary driver mutation, such as EGFR, ALK, ROS1, NTRK, or BRAF, the patient must be treated with the appropriate targeted therapy first. Patient is eligible if RET fusion is confirmed AND patient has undergone initial therapy for his/her driver mutation, or

1b. Pathologically documented and definitively diagnosed RET mutation in advanced MTC patients who are treatment naïve or who have been previously treated with MKI therapy, or

1c. Pathologically documented and definitively diagnosed advanced solid tumor with an oncogenic RET fusion previously treated with standard of care appropriate for the tumor type.

2. If previously treated with a selective RET inhibitor (e.g., RETEVMO), confirm patient has not progressed but has discontinued due to adverse event(s).

3. Patient is not eligible for an ongoing study of pralsetinib or cannot access an ongoing study of pralsetinib.

4. Patient is ≥ 12 years of age. 5. Patient has adequate vital organ function, including heart, lungs, liver, kidneys, bone marrow and endocrine, and is expected to tolerate therapy with a tyrosine kinase inhibitor.

6. No presence of clinically symptomatic interstitial lung disease or interstitial pneumonitis, including radiation pneumonitis (i.e., affecting activities of daily living or requiring therapeutic intervention).

7. Patient or patient's legal guardian, if permitted by local regulatory authorities, intends to provide informed consent prior to the start of treatment with pralsetinib.

8. Patient does not require therapy with a concomitant medication that is a strong inhibitor or strong inducer of cytochrome P450 (CYP) 3A4.

9. Patient has not received treatment with any systemic anticancer therapy (except for immunotherapy or other antibody therapies) and all forms of radiotherapy within 14 days or 5 half-lives prior to the first dose of pralsetinib. Pralsetinib may be started within these washout periods if considered by the healthcare provider to be safe and within the best interest of the patient, with prior Sponsor approval.

10. Patient has not received treatment with any immunotherapy or other antibody therapy within 28 days prior to the first dose of pralsetinib (immune related toxicities must have resolved to < Grade 2 prior to starting pralsetinib).

11. Patient has not had a major surgical procedure (minor surgical procedures such as central venous catheter placement, tumor needle biopsy, and feeding tube placement are not considered major surgical procedures) within 14 days prior to the first dose of pralsetinib.

12. Women must be willing, if not postmenopausal or surgically sterile, to abstain from sexual intercourse or employ highly effective contraception during pralsetinib administration period and for at least 30 days after the last dose of pralsetinib. Men, if not surgically sterile, must be willing to abstain from sexual intercourse or employ highly effective contraception during pralsetinib administration period and for at least 90 days after the last dose of pralsetinib.

13. Women must not be pregnant or breastfeeding.

Min Age: 12 Years | Sex: All
Age Groups: Child, Adult, Older Adult